CLINICAL TRIAL: NCT04796662
Title: CT Lucia 601 IOL Implantation in the Sulcus
Acronym: CLUS
Status: Terminated | Type: Observational
Why Stopped: Poor recruitment
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S64878
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Cataract; Complicata; Posterior Capsule Tear; Lens Dislocation
Keywords: CT Lucia 601 lens
MeSH Terms: conditions — Cataract; Lens Subluxation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To perform a retrospective investigation of the CT Lucia 601 IOL implantation in the sulcus

DETAILED DESCRIPTION:
The purpose of the study is to collect data that are parameters of post-IOL implantation safety:

* Questionnaire on subjective quality of vision
* Centration and anteroposterior position of the IOL (using biometry)
* Presence and quantification of any inflammation or pigment present in the anterior chamber (flare meter)
* Refractive outcome, with calculation of customized A-constant of the CT Lucia 601 IOL in-the-sulcus and quantification of higher-order aberrations (HOA)
* General safety-parameters:

  * Visual acuity
  * Intra-ocular pressure
  * Presence of macular edema or retinal nerve fiber layer (RNFL) thinning (SD-OCT)
  * Any adverse ophthalmic events

ELIGIBILITY:
Inclusion Criteria:

* Patients with an implantation of a CT Lucia 601 lens for different reasons:

  * During vitrectomy to treat a complicated cataract surgery and had the implantation of a CT Lucia 601 IOL in the sulcus or patients
  * During phaco surgery with a posterior capsule tear that necessitated the implantation of the implant lens in the sulcus
  * Explantation of an in-the-bag lens and implantation of a CT Lucia 601 as replacement lens (e.g. to treat opacification of the implant lens or intolerance of the implant lens).
* Age : > 18 years
* Signed informed consent
* Preoperative myopia less than 10 diopters
* Implantation of the CT Lucia IOL at least six months earlier

Exclusion Criteria:

* History of uveitis
* Ocular pathology or history that could influence the biometry of the effective lens position, such as ocular trauma with zonulolysis, congenital iris- or lens defects etc.
* Any eye condition influencing the lens position (to be specified) according to the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who had an implantation of the CT Lucia 601 lens
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
safety of the CT Lucia 601 IOL in the sulcus | 2019-2020
  determine whether the CT Lucia 601 IOL can be used safely in the sulcus

CONTACTS AND LOCATIONS:
Overall Officials: Peter Stalmans, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams Brabant, Belgium

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT04796662/Prot_SAP_000.pdf